CLINICAL TRIAL: NCT01309750
Title: Small Bowel Transit Time in Clostridium Difficile Colitis
Status: Terminated | Type: Observational
Why Stopped: logistics
Sponsor: Corewell Health East (Other)
Responsible Party: Sponsor
Other Study IDs: 2011-008
Record Dates: First submitted 2011-03-03; First posted 2011-03-07 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2012-09

CONDITIONS: Clostridium Difficile Colitis
MeSH Terms: conditions — Enterocolitis, Pseudomembranous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- C. diff: Patients with Clostridium difficile colitis admitted to the intensive care unit will be the study group.
  Interventions: Radiation: Small Bowel Transit Study

INTERVENTIONS:
Radiation: Small Bowel Transit Study — Patients that are enrolled and consented in the study will be given 300ml of water containing 5 millicurie (mCi) of technetium-99m (Tc-99m) diethylenetriamine pentaacetate (DTPA). This nuclear tracer/water mix will either be drank orally or placed down a nasogastric tube to begin the study. The patient will have to have nothing else to eat or drink for the duration of the study. The patients will have a nuclear scan performed at 2, 4, and 6 hours after ingestion of the nuclear tracer.

SUMMARY:
Clostridium difficile is a bacteria that can infect the colon and cause severe diarrhea in patients after recent antibiotic use. The current standard of care treatment for severe C. diff. consists of oral vancomycin and/or intravenous metronidazole. When treatment is unsuccessful, it can lead to need for removal of the entire colon or even death. In fact, mortality rates in the literature range from 11-37% for C. diff. The most commonly quoted mortality rate is 14% for severe infection. It is believed that the failure of treatment may stem from an adynamic ileus (paralysis of the small bowel). This ileus may prevent the oral vancomycin from reaching the colon and therefore it does not treat the problem. Vancomycin functions by direct contact with the colon. It is presumed that this paralysis of the small intestine is present but has never been proven. The objective of the study is to prove that there is an adynamic ileus present in c. diff colitis and therefore lead to investigations into improved treatment.

DETAILED DESCRIPTION:
Patients in the intensive care unit are eligible to participate in the study A pregnancy test will be checked if applicable. Patients that are enrolled and consented in the study will be given 300ml of water containing 5 millicurie (mCi) of technetium-99m (Tc-99m) diethylenetriamine pentaacetate (DTPA). This nuclear tracer/water mix will either be drank orally or placed down a nasogastric tube to begin the study. The patient will have to have nothing else to eat or drink for the duration of the study. The patients will have a nuclear scan performed at 2, 4, and 6 hours after ingestion of the nuclear tracer. The images at 2 and 6 hours will be taken in the nuclear medicine department while the 4 hour image will be taken in the ICU. The 2 and 6 hour studies must be conducted in the nuclear medicine department to allow for special equipment to be used. This equipment is necessary to allow for computer calculation to be made. The 4 hour scan is to check for progress of the tracer and does not require calculations/measurements. Therefore, a mobile scanner can be utilized. The image will be taken for 60 seconds. The images obtained will then be interpreted by the nuclear medicine department to determine the transit time of the tracer from the stomach to the terminal ileum and cecum. The data obtained from the subjects will be compare to previously obtained data for normal subjects. A normal study has been defined as 40% of the tracer reaching the terminal ileum by 6 hours. Any time longer than 6 hours is deemed an abnormal study with delayed small bowel transit time.

ELIGIBILITY:
Inclusion Criteria:

* ICU patient
* positive c. diff PCR or visualization of pseudomembranes on colonoscopy
* able to give consent or have representative to give consent
* ability to drink contrast or have a previously placed nasogastric tube
* approval from the intensivist on duty/ICU Attending physician

Exclusion Criteria:

* Under age 18
* pregnant
* need for gastric motility medications
* need for anti-diarrheal medication
* need for surgery
* previous small bowel or gastric surgery
* inability to drink nuclear tracer without nasogastric tube in place
* hypotension requiring vasoactive agents
* APACHE II score greater than 30

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with clostridium difficile colitis.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2011-04; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc B Grodsky, Principal Investigator — Corewell Health East
Locations (1):
- William Beaumont Hospital, Royal Oak, Michigan, United States